CLINICAL TRIAL: NCT02354079
Title: HYPOCHOL : A Genetically-based Strategy to Identify New Targets in Cholesterol Metabolism
Acronym: HYPOCHOL
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RC14_0400
Record Dates: First submitted 2015-01-14; First posted 2015-02-03 (Estimated); Last update posted 2023-08-04 (Actual); Status verified 2023-08

CONDITIONS: Hypobetalipoproteinemia
Keywords: Low LDL-C; Target Identification; Genetic; Endocrinology; Cardiovascular Disease
MeSH Terms: conditions — Hypobetalipoproteinemias; Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- genetic analysis (Other)
  Interventions: Genetic: hypobetalipoproteinemia genetic and genotypic screening

INTERVENTIONS:
Genetic: hypobetalipoproteinemia genetic and genotypic screening

SUMMARY:
The aim of this study is to identify new targets in cholesterol metabolism thanks to a genetically-based strategy.

DETAILED DESCRIPTION:
The goal is to recruit 400 subjects: 200 adult subjects with familial hypobetalipoproteinemia (FHBL) (index cases) plus 200 additional related subjects in at least 10 large informative FHBL families, in which there is no known mutation in FHBL genes.

The patient care is modified: patient will have an Hospital Anxiety and Depression (HAD) questionnaire (focus on depressive syndrome), a food diary, and some additional blood analysis (including genetic analysis).

One of the main issue to recruit FHBL patients is the fact that they are asymptomatic and that FHBL is not identified as a serious illness by their general physicians.

Step-1. Excluding mutations in selected candidate genes As a first approach to screen candidate genes and exclude patients with known mutations, the investigators developed a custom design based on the Haloplex™ technology (Agilent® Technologies) to perform high-throughput sequencing of the coding regions of 10 genes, including those previously described in FHBL (apolipoprotein B (APOB), Proprotein convertase subtilisin/kexin type 9 (PCSK9)), Microsomal triglyceride transfer protein (MTP or ABL), chylomicron retention disease (CMRD), Secretion associated, Ras related GTPase (SARA2 gene), as well as 6 additional candidate genes in cholesterol metabolism (low density lipoprotein receptor (LDLR), Sortilin (SORT1), Inducible Degrader of the LDL receptor (IDOL), Cholesteryl ester transfer protein (CETP), Apolipoprotein E (ApoE) and Angiopoietin-like Protein 3 (ANGTPL3)). All the recruited index cases (n=200) will be genotyped to select only those without mutations in previously described genes, being approximately 50% of our index case cohort.

Step-2. Identification of informative families and exome sequencing In patients without identified mutations, the investigators will conduct a familial screening in order to identify other cases of FHBL among proband relatives. An analysis of fasting plasma lipid parameters (total cholesterol (TC), High density lipoprotein cholesterol (HDL-C), Low-Density Lipoproteins (LDL-C) and triglycerides (TG)) will be performed for each related. Affected subjects will be determined by a spontaneous LDL-C < 80 mg/dl and/or apoB < 50 mg/dl. In contrast, non-affected subjects will display LDL-C > 80 mg/dl and/or apoB > 50 mg/dl.

For large families, the investigators will then combine whole-exome sequencing and linkage analysis to identify any novel genetic variant likely explaining FHBL. Depending on family pedigree, whole-exome sequencing (WES) will be performed on 2 to 5 patients per family. All relatives will be genotyped for linkage analysis.

In parallel to this genetic approach, a regional epidemiological analysis will be performed to identify some geographical clusters with a high prevalence of the disease, as developed in the project named VaCaRMe (for Vascular and Cardiac, Respiratory and Metabolic overcome diseases)

An additional aim, based on an exhaustive phenotyping of FHBL patients, is to investigate the safety of very low LDL-C and to perform some genotype-phenotype correlations in patients with FHBL population."

ELIGIBILITY:
Inclusion Criteria:

* For index cases without family screening:

  o Patient with HBL: fasting LDL-C ≤ 50 mg/dl.
* For familial affected cases:

  * Relative with HBL: fasting LDL-C ≤ 80 mg/dl and/or Apo B ≤ 50 mg/dl and at least one related family case suffering from HBL.

All subjects, including familial non-affected cases, must give written consent (dated and signed) to participate at the constitution of biobank (including DNA samples and urine samples).

Exclusion Criteria:

* Use of lipid-lowering drugs (statins, fibrates, ezetimibe, bile-acid sequestering resin) or nutraceuticals known to affect lipids (red yeast rice, margarine and dairy with plant sterol)
* Patient screened within an extreme metabolic disturbance (emergency situations, sepsis, hospitalization in intensive care unit)
* Patients with hyperthyroidism, severe liver failure, end stage chronic kidney disease, serious pancreatic failure, anemia related to thalassemia or sickle cell disease, strict vegan diet or malnutrition
* Refusal of the patient or his legal representative to participate in the study"

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 435 (Actual)
Dates: Start 2016-01-07 (Actual); Primary Completion 2022-01-07 (Actual); Study Completion 2032-01-07 (Estimated)

PRIMARY OUTCOMES:
type and number of genetic abnormalities leading to FHBL | ten years
  To identify new gene involved in FHBL and determine genetic cause of FHBL (Patients with FHBL and their relatives will be recruited to establish familial forms of FHBL in large informative families with no mutations in known classical FHBL genes. This will allow perform genetic analysis using new approaches to genetic broadband (exome sequencing analysis + linkage analysis). This approach will allow specify which chromosomal regions are shared only by affected individuals, and identify new candidate genes).

OTHER OUTCOMES:
number of phenotypes associated to genotype of FHBL and very low LDL-C | ten years
  To determine number of phenotypes associated to genotype of FHBL and very low LDL-C. (Liver steatosis, Glucose homeostasis, Cancer, Depression scores, Cardiovascular diseases).

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte AUTHIER, Doctor, Principal Investigator — Health Care Centers of French Health Insurance in Saint-Nazaire; Didier GOXE, Principal Investigator — Health Care Centers of French Health Insurance in La Roche sur Yon
Locations (1):
- CHU de Nantes, Nantes, France